CLINICAL TRIAL: NCT02854397
Title: Determination of Specific Biomarkers of Acute Attack of Angioedema Within Pediatric Population
Acronym: BRADYKID
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC15.180
Record Dates: First submitted 2016-07-18; First posted 2016-08-03 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Hereditary Angioedema; Healthy Volunteers
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with hereditary angioedema: A blood sample will be performed in crisis and 7 days after the crisis.
  Interventions: Other: blood sample
- patients with angioedema resulting of mast cell activation: A blood sample will be performed in crisis and 7 days after the crisis.
  Interventions: Other: blood sample
- healthy patients, without angioedema: A quantity of additional blood was taken from eligible patients who had a scheduled blood sample.
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
In emergency room, this is crucial to diagnose an acute attack of hereditary angioedema (HAE) to quickly provide the efficient treatment. Currently, there is no specific biomarker for acute attack of bradykinin-mediated angioedema to help clinicians for patient care. However, previous works are carried out for that purpose. All the potential candidate biomarkers must be validated in prospective studies to estimate their specificity and sensitivity values, and to understand their potential utility in patient care.

The main goal of this clinical trial is to estimate the diagnostic value of VE-cadherin in pediatric population, for the differential diagnosis between HAE crisis and angioedema resulting of mast cell activation crisis (the main differential diagnosis of HAE).

ELIGIBILITY:
Inclusion Criteria:

For HAE: patient with a documented diagnosis of HAE:

* type I (from an antigenic deficiency of the C1 esterase inhibitor) or type II (from a functional deficiency of the C1 esterase inhibitor). The existence of a mutation in SERPING1 was not necessary for the inclusion
* HAE with normal C1-INH (ex type III) with a required mutation in FXII gene or with a typical family history of HAE diagnosed by a specialized physician belonging to CREAK network.

For AE resulting of mast cell activation: a documented diagnosis of AE resulting of mast cell activation included:

* mastocytosis,
* chronic spontaneous urticaria,
* acute urticaria after exposure of allergen during allergy challenge tests,
* mast cell activation syndrome.

For the control group:

* composed of patients who presented a stabilized disease (that was not infectious, not auto-inflammatory or inflammatory disease and without implication of endothelial cells).

Exclusion Criteria:

* Over 18 years or under 1 year.
* Diagnosis of HAE with a normal C1 esterase inhibitor or AE of unknown aetiology.
* Patients with HAE who received an acute attack treatment before the blood sample (the C1 esterase inhibitor concentrate or a bradykinin B2 receptor antagonist); patients with HAE who received a prophylactic treatment (danazol).
* Patients who were treated by omalizumab or corticosteroid treatment.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with hereditary angioedema patients with angioedema resulting of mast cell activation healthy patients, without angioedema
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
VE-cadherin level | Half a day
  For the diagnosis of acute attack of hereditary angioedema

SECONDARY OUTCOMES:
Dosage of VE-cadherin (vascular endothelial) | Half a day
  Analysis of the cleaved fragments from high molecular weight kininogen
Dosage of Fc KHPM | Half a day
  Analysis of the cleaved fragments from high molecular weight kininogen
Dosage of D-dimer | Half a day
  Analysis of the cleaved fragments from high molecular weight kininogen
Dosage of Tryptase | Half a day
  Analysis of the cleaved fragments from high molecular weight kininogen

CONTACTS AND LOCATIONS:
Overall Officials: Anne Pagnier, Principal Investigator — University Hospital, Grenoble
Locations (14):
- France (14):
  - University hospital angers, Angers
  - University Hospital Besançon, Besançon
  - University hospital Bordeaux, Bordeaux
  - University hopital Clermont-Ferrand, Clermont-Ferrand
  - University Hospital Grenoble, Grenoble
  - University Hospital Lille, Lille
  - University Hospital Lyon, Lyon
  - University hospital Marseille, Marseille
  - University hospital Montpellier, Montpellier
  - University hospital Nancy, Nancy
  - General Hospital, Niort
  - university hospital Saint-Antoine (AP-HP), Paris
  - University hospital Rouen, Rouen
  - University hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boccon-Gibod I, Bouillet L. [Angioedema and urticaria]. Ann Dermatol Venereol. 2014 Nov;141 Suppl 3:S586-95. doi: 10.1016/S0151-9638(14)70162-0. French. PMID 25539680
- [Background] Pagnier A. [Hereditary angioedema in childhood. Diagnosis and therapeutic challenges]. Presse Med. 2015 Jan;44(1):89-95. doi: 10.1016/j.lpm.2014.07.018. Epub 2014 Dec 12. French. PMID 25511651
- [Background] Dinkel HP, Maroske J, Schrod L. Sonographic appearances of the abdominal manifestations of hereditary angioedema. Pediatr Radiol. 2001 Apr;31(4):296-8. doi: 10.1007/s002470000409. PMID 11321752
- [Background] Bygum A. Hereditary angio-oedema in Denmark: a nationwide survey. Br J Dermatol. 2009 Nov;161(5):1153-8. doi: 10.1111/j.1365-2133.2009.09366.x. Epub 2009 Jun 22. PMID 19709101
- [Background] Farkas H. Pediatric hereditary angioedema due to C1-inhibitor deficiency. Allergy Asthma Clin Immunol. 2010 Jul 28;6(1):18. doi: 10.1186/1710-1492-6-18. PMID 20667121
- [Background] El-Hachem C, Amiour M, Guillot M, Laurent J. [Hereditary angioneurotic edema: a case report in a 3-year-old child]. Arch Pediatr. 2005 Aug;12(8):1232-6. doi: 10.1016/j.arcped.2005.03.052. French. PMID 15890504
- [Background] Farkas H. Management of upper airway edema caused by hereditary angioedema. Allergy Asthma Clin Immunol. 2010 Jul 28;6(1):19. doi: 10.1186/1710-1492-6-19. PMID 20667122
- [Background] Sanchez A, Ecochard A, Maestracci M, Rodiere M. [Hereditary angioedema causing colocolic intussusception]. Arch Pediatr. 2008 Mar;15(3):271-4. doi: 10.1016/j.arcped.2007.12.004. Epub 2008 Mar 10. French. PMID 18329867
- [Background] Pritzker HA, Levin TL, Weinberg G. Recurrent colocolic intussusception in a child with hereditary angioneurotic edema: reduction by air enema. J Pediatr Surg. 2004 Jul;39(7):1144-6. doi: 10.1016/j.jpedsurg.2004.03.075. PMID 15213920
- [Background] Parisi G, Chiarelli A, Squadrone NP, Galante E. Hereditary angioedema, a rare cause of recurrent abdominal pain. A report of 2 clinical cases and comments of a general nature Allergy Asthma Proc. 2013 Jul-Aug;34(4):312-27
- [Background] MacGinnitie AJ. Pediatric hereditary angioedema. Pediatr Allergy Immunol. 2014 Aug;25(5):420-7. doi: 10.1111/pai.12168. Epub 2013 Dec 9. PMID 24313851
- [Background] Deroux A, Vilgrain I, Dumestre-Perard C, Boccon-Gibod I, Bouillet L. Towards a specific marker for acute bradykinin-mediated angioedema attacks: a literature review. Eur J Dermatol. 2015 Jul-Aug;25(4):290-5. doi: 10.1684/ejd.2015.2547. PMID 25905454
- [Background] Cugno M, Zanichelli A, Bellatorre AG, Griffini S, Cicardi M. Plasma biomarkers of acute attacks in patients with angioedema due to C1-inhibitor deficiency. Allergy. 2009 Feb;64(2):254-7. doi: 10.1111/j.1398-9995.2008.01859.x. Epub 2008 Dec 4. PMID 19076541
- [Background] Hogan AD, Schwartz LB. Markers of mast cell degranulation. Methods. 1997 Sep;13(1):43-52. doi: 10.1006/meth.1997.0494. PMID 9281467
- [Background] Brickman CM, Frank MM, Kaliner M. Urine-histamine levels in patients with hereditary angioedema (HAE). J Allergy Clin Immunol. 1988 Sep;82(3 Pt 1):403-6. doi: 10.1016/0091-6749(88)90012-7. PMID 3170987
- [Background] Payne V, Kam PC. Mast cell tryptase: a review of its physiology and clinical significance. Anaesthesia. 2004 Jul;59(7):695-703. doi: 10.1111/j.1365-2044.2004.03757.x. PMID 15200544
- [Background] Kasperska-Zajac A, Grzanka A, Czecior E, Misiolek M, Rogala B, Machura E. Acute phase inflammatory markers in patients with non-steroidal anti-inflammatory drugs (NSAIDs)-induced acute urticaria/angioedema and after aspirin challenge. J Eur Acad Dermatol Venereol. 2013 Aug;27(8):1048-52. doi: 10.1111/j.1468-3083.2012.04486.x. Epub 2012 Feb 21. PMID 22348297
- [Background] Fujii K, Konishi K, Kanno Y, Ohgou N. Acute urticaria with elevated circulating interleukin-6 is resistant to anti-histamine treatment. J Dermatol. 2001 May;28(5):248-50. doi: 10.1111/j.1346-8138.2001.tb00126.x. PMID 11436361
- [Background] Kasperska-Zajac A, Brzoza Z. Increased D-dimer concentration in plasma of patients with severe acute urticaria. Br J Dermatol. 2009 Dec;161(6):1409-10. doi: 10.1111/j.1365-2133.2009.09466.x. Epub 2009 Sep 15. No abstract available. PMID 19754863
- [Background] Brevet: w/o 2008 062314 circulating ve-cadherin as a predictive marker of sensitivity or resistance to anti-tumoral treatment, and improved method for the detection of soluble proteins.
- [Background] Bouillet L, Sidibe A, Polena H, Mannic T, Deroux A, Stidder B, Vittecoq O, Vilgrain I. [Endothelial junctions: exploiting their instability in the development of biomarkers for vascular remodelling]. Med Sci (Paris). 2014 Jun-Jul;30(6-7):633-5. doi: 10.1051/medsci/20143006012. Epub 2014 Jul 11. No abstract available. French. PMID 25014453
- [Background] Bouillet L, Vilgrain I. VE-cadherin, a potential marker for endothelial cell activation during hereditary angioedema attacks. J Allergy Clin Immunol. 2014 Jul;134(1):241. doi: 10.1016/j.jaci.2014.04.016. Epub 2014 May 27. No abstract available. PMID 24875615
- [Background] Sidibe A, Polena H, Pernet-Gallay K, Razanajatovo J, Mannic T, Chaumontel N, Bama S, Marechal I, Huber P, Gulino-Debrac D, Bouillet L, Vilgrain I. VE-cadherin Y685F knock-in mouse is sensitive to vascular permeability in recurrent angiogenic organs. Am J Physiol Heart Circ Physiol. 2014 Aug 1;307(3):H455-63. doi: 10.1152/ajpheart.00774.2013. Epub 2014 May 23. PMID 24858856
- [Background] Sidibe A, Polena H, Razanajatovo J, Mannic T, Chaumontel N, Bama S, Marechal I, Huber P, Gulino-Debrac D, Bouillet L, Vilgrain I. Dynamic phosphorylation of VE-cadherin Y685 throughout mouse estrous cycle in ovary and uterus. Am J Physiol Heart Circ Physiol. 2014 Aug 1;307(3):H448-54. doi: 10.1152/ajpheart.00773.2013. Epub 2014 May 23. PMID 24858855
- [Background] Bouillet L, Mannic T, Arboleas M, Subileau M, Massot C, Drouet C, Huber P, Vilgrain I. Hereditary angioedema: key role for kallikrein and bradykinin in vascular endothelial-cadherin cleavage and edema formation. J Allergy Clin Immunol. 2011 Jul;128(1):232-4. doi: 10.1016/j.jaci.2011.02.017. Epub 2011 Mar 24. No abstract available. PMID 21439626
- [Background] Suffritti C, Zanichelli A, Maggioni L, Bonanni E, Cugno M, Cicardi M. High-molecular-weight kininogen cleavage correlates with disease states in the bradykinin-mediated angioedema due to hereditary C1-inhibitor deficiency. Clin Exp Allergy. 2014 Dec;44(12):1503-14. doi: 10.1111/cea.12293. PMID 24552232
- [Background] Kahn R, Herwald H, Muller-Esterl W, Schmitt R, Sjogren AC, Truedsson L, Karpman D. Contact-system activation in children with vasculitis. Lancet. 2002 Aug 17;360(9332):535-41. doi: 10.1016/S0140-6736(02)09743-X. PMID 12241658
- [Background] Ghannam A, Sellier P, Defendi F, Favier B, Charignon D, Lopez-Lera A, Lopez-Trascasa M, Ponard D, Drouet C. C1 inhibitor function using contact-phase proteases as target: evaluation of an innovative assay. Allergy. 2015 Sep;70(9):1103-11. doi: 10.1111/all.12657. Epub 2015 Jun 9. PMID 26010015
- [Background] Adam SS, Key NS, Greenberg CS. D-dimer antigen: current concepts and future prospects. Blood. 2009 Mar 26;113(13):2878-87. doi: 10.1182/blood-2008-06-165845. Epub 2008 Nov 13. PMID 19008457
- [Background] Blohme G. Treatment of hereditary angioneurotic oedema with tranexamic acid. A random double-blind cross-over study. Acta Med Scand. 1972 Oct;192(4):293-8. doi: 10.1111/j.0954-6820.1972.tb04818.x. No abstract available. PMID 4562897
- [Background] Brown NJ, Gainer JV, Stein CM, Vaughan DE. Bradykinin stimulates tissue plasminogen activator release in human vasculature. Hypertension. 1999 Jun;33(6):1431-5. doi: 10.1161/01.hyp.33.6.1431. PMID 10373228
- [Background] Cugno M, Hack CE, de Boer JP, Eerenberg AJ, Agostoni A, Cicardi M. Generation of plasmin during acute attacks of hereditary angioedema. J Lab Clin Med. 1993 Jan;121(1):38-43. PMID 8426080
- [Background] Frank MM, Sergent JS, Kane MA, Alling DW. Epsilon aminocaproic acid therapy of hereditary angioneurotic edema. A double-blind study. N Engl J Med. 1972 Apr 13;286(15):808-12. doi: 10.1056/NEJM197204132861503. No abstract available. PMID 4551861
- [Background] Joseph K, Tholanikunnel BG, Wolf B, Bork K, Kaplan AP. Deficiency of plasminogen activator inhibitor 2 in plasma of patients with hereditary angioedema with normal C1 inhibitor levels. J Allergy Clin Immunol. 2016 Jun;137(6):1822-1829.e1. doi: 10.1016/j.jaci.2015.07.041. Epub 2015 Sep 26. PMID 26395818
- [Background] Kaplan AP, Austen KF. A prealbumin activator of prekallikrein. II. Derivation of activators of prekallikrein from active Hageman factor by digestion with plasmin. J Exp Med. 1971 Apr 1;133(4):696-712. doi: 10.1084/jem.133.4.696. PMID 4251126
- [Background] Kleniewski J, Blankenship DT, Cardin AD, Donaldson V. Mechanism of enhanced kinin release from high molecular weight kininogen by plasma kallikrein after its exposure to plasmin. J Lab Clin Med. 1992 Jul;120(1):129-39. PMID 1535355
- [Background] Kluft C, Trumpi-Kalshoven MM, Jie AF, Veldhuyzen-Stolk EC. Factor XII-dependent fibrinolysis: a double function of plasma kallikrein and the occurrence of a previously undescribed factor XII- and kallikrein-dependent plasminogen proactivator. Thromb Haemost. 1979 Jun 30;41(4):756-73. PMID 483248
- [Background] Nielsen EW, Johansen HT, Hogasen K, Wuillemin W, Hack CE, Mollnes TE. Activation of the complement, coagulation, fibrinolytic and kallikrein-kinin systems during attacks of hereditary angioedema. Scand J Immunol. 1996 Aug;44(2):185-92. doi: 10.1046/j.1365-3083.1996.d01-298.x. PMID 8711433
- [Background] Reshef A, Zanichelli A, Longhurst H, Relan A, Hack CE. Elevated D-dimers in attacks of hereditary angioedema are not associated with increased thrombotic risk. Allergy. 2015 May;70(5):506-13. doi: 10.1111/all.12587. Epub 2015 Feb 23. PMID 25640891